CLINICAL TRIAL: NCT04114240
Title: French Study in Real Life Evaluating Xybilun: Convenience and Erection Induction Related to a New Administration in Orodispersible Film
Brief Title: French Study in Real Life Evaluating Xybilun
Acronym: XY-FILM
Status: Completed | Type: Observational
Sponsor: Laboratoires Genévrier (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-A03204-49
Record Dates: First submitted 2018-09-06; First posted 2019-10-03 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Erectile Dysfunction
Keywords: erectil dysfunction; sildenafil; xybilun
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Xybilun: mild erectil dysfunction: Patient who has never been treated for his ED (erectil dysfunction), with mild ED (score IIEF-6 between 22 and 25) and begin treatment at 50 mg
  Interventions: Drug: Xybilun
- Xybilun: moderate erectil dysfunction: Patient who has never been treated for his ED (erectil dysfunction), with moderate ED (score IIEF-6 between 11 and 21) and begin treatment at 50 mg
  Interventions: Drug: Xybilun
- Xybilun: severe erectil dysfunction: Patient who has never been treated for his ED (erectil dysfunction), with severe ED (score between 6 and 10) and begin treatment at 50 mg
  Interventions: Drug: Xybilun
- Xybilun switch: Substitution dose to dose of previous treatment by Xybilun whatever the severity of ED.
  Interventions: Drug: Xybilun

INTERVENTIONS:
Drug: Xybilun — Erectil dysfunction, Viagra generic (sildénafil)

SUMMARY:
Collecting Xybilun (Viagra's generic) efficacity, tolerance, convenience and patients/doctors satisfaction's data at different doses (50-75-100 mg), is the aim of the study.

DETAILED DESCRIPTION:
Study design

Population Patients without prior treatment with a first Xybilun prescription Patients already treated for who the treatment is remplaced by Xybilun

Study perimeter 400 patients 50 investigators (sexologists, urologists)

ELIGIBILITY:
Inclusion Criteria:

* Age > or equal 18 years
* Erectile dysfunction at V1 light (group 1), moderate (group 2), severe (group 3): IIEF-6 score between 6 and 25 (IIEF-6 questions 1-5 and question 15)
* More than 3 sexual intercourse
* First prescription of Xybilun (gr 1,2,3) or subtitution (gr 4)
* Information and non-opposition

Exclusion Criteria:

* Sildénafil hypersensitivity
* Treatment with nitrogen oxide or guanylate cyclase
* Patient with sexual intercourse prohibited
* NOIANA
* Alpha-blocker during past 3 months
* Norvir
* Participation in an other clinical trial
* Patient unable to read properly an information sheet
* Patient under guardianship/curatorship

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Man suffering from all type of erectil dysfunction (light, moderate, severe).
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-04-26 (Actual)

PRIMARY OUTCOMES:
Patients who has never been treated for ED (group 1,2,3) : responder patients rate at V3 (IIEF-6 : international index of erectil function) | 3 months
  Group 1: patient good responder if there is an increase of at least 2 points regarding score of IIEF-6; Group 2: patient good responder if there is an increase of at least 5 points regarding score of IIEF-6; Group 3: patient good responder if there is an increase of at least 7 points regarding score of IIEF-6;
Patients with treatment substitution (group 4): satisfaction of Xybilun vs previous treatment at V3 (Likert scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied) | 3 months
  Likert scale in 5 point evaluated at V3: "Are you more satisfied regarding you previous treatment then your current treatment?" Patient improved if his answer is "satisfied" (score 4) or "very satisfied" (score 5).

SECONDARY OUTCOMES:
Patients who has never been treated for ED (group 1,2,3) : responder patients at V2 Month 1 (IIEF-6) | 1 month
  score IIEF-6 (international index erectif function) score frome 0 to 30 : 22-25 ED mild, 11-21 ED moderate, 6-10 ED severe Group 1: patient good responder if there is an increase of at least 2 points regarding score of IIEF-6; Group 2: patient good responder if there is an increase of at least 5 points regarding score of IIEF-6; Group 3: patient good responder if there is an increase of at least 7 points regarding score of IIEF-6;
Patients who has never been treated for ED (group 1,2,3) : overall satisfaction at 1 month and 3 month | 1 month and 3 months
  GAQ Global Assessment Questionnaire : 1 question "does the treatment has ameliorate your erection" Y/N
Patients who has never been treated for ED (group 1,2,3) : Patient Xybilun and investigator satisfaction at V2 month 1 and V3 month 3 | 1 month and 3 months
  Likert scale (5 points) : 1 question : "are you satisfied of Xybilun?" (Likert scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied)
Patients who has never been treated for ED (group 1,2,3) : convenience at V2 month 1 and V3 month 3 (Likert scale) | 1 month and 3 months
  Likert scale (5 points) : 1 question "How convenient Xybilun is ?) (Likert scale 5 points : 1-Not convenient at all, 2-not very convenient, 3-nor convenient nor unconvenient, 4- convenient, 5-very convenient)
Patients who has never been treated for ED (group 1,2,3) : Partner satisfaction (Likert scale) at month 3 | 3 months
  Likert scale (5 points): (optional data) 1 question : "are you satisfied of Xybilun?" (Likert scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied)
Patients with treatment substitution (group 4): International index of erectile function (IIEF) evolution (IIEF15) | 1 month and 3 months
  IIEF15 international index of erectile function (15 questions scored from 0 to 5) ; score from 0 to 75 to evaluate globale erectil dysfunction (not used for classify the disfunction only to see the score evolution in the time)
Patients with treatment substitution (group 4): satisfaction (patient/investigator) of previous treatment evaluated at V1 (Day 0) (Likert scale) | Day 0
  Likert scale (5 points) : "Are you more satisfied regarding you previous treatment then your current treatment?" scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied)
Patients with treatment substitution (group 4): satisfaction of Xybilun (patient/investigator) at V2 month 1 and V3 month 3 (Likert scale) | 1 month and 3 months
  Likert scale (5 points) : 1 question : "are you satisfied of Xybilun?" (Likert scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied)
Patients with treatment substitution (group 4): convenience previous treatment at V1 (day 0) (Likert scale) | Day 0
  Likert scale (5 points) 1 question "How convenient you previous treatment was ?) (Likert scale 5 points : 1-Not convenient at all, 2-not very convenient, 3-nor convenient nor unconvenient, 4- convenient, 5-very convenient)
Patients with treatment substitution (group 4): convenience Xybilun (patient) at V2 month 1 and V3 month 3 (Likert scale) | 1 month and 3 months
  Likert scale (5 points) 1 question "How convenient Xybilun is ?) (Likert scale 5 points : 1-Not convenient at all, 2-not very convenient, 3-nor convenient nor unconvenient, 4- convenient, 5-very convenient)
Patients with treatment substitution (group 4): Partner satisfaction at V3 month 3 (Likert scale) | 3 months
  ikert scale (5 points): (optional data) 1 question : "are you satisfied of Xybilun?" (Likert scale 5 points : 1-Not satisfied at all, 2-not very satisfied, 3-nor satisfied nor unsatisfied, 4- satisfied, 5-very satisfied)
Patients with treatment substitution (group 4): reasons of treatment substitution | Day 0
  1 question : "reason of substitution : lack of efficacy, adverse event, bad taste, difficulty of taking, price elevated, ED healing, other (precise)"
Patients with treatment substitution (group 4): efficacy of Xybilun comparing score IIEF-6 before/after treatment | 1 month and 3 months
  score IIEF-6 (international index erectif function) score frome 0 to 30 : 22-25 ED mild, 11-21 ED moderate, 6-10 ED severe ED mild: responder if there is an increase of at least 2 points regarding score of IIEF-6; ED moderate: responder if there is an increase of at least 5 points regarding score of IIEF-6; ED severe: responder if there is an increase of at least 7 points regarding score of IIEF-6;
safety | 1 month and 3 months
  Adverse event : description of AE : open field, related or not to Xybilun, gravity scale (mild, moderate, severe, healththreatening)

CONTACTS AND LOCATIONS:
Overall Officials: DROUPY SD Stéphane, Urologist, Principal Investigator — CHU Nîmes
Locations (1):
- CHU Nîmes, Nantes, Haute-Bretagne, France